CLINICAL TRIAL: NCT02851134
Title: Search for New Genetic Mutations Major Effect in Crohn's Disease
Acronym: MC-WES
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2013_53; 2014-A00023-44 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2016-06-07; First posted 2016-08-01 (Estimated); Last update posted 2019-02-28 (Actual); Status verified 2019-02

CONDITIONS: Crohn Disease
Keywords: genetic
MeSH Terms: conditions — Crohn Disease | interventions — Genetic Testing; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples stools samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Crohn disease subject: Crohn disease affected subject
  Interventions: Genetic: genetic analysis; Biological: blood and stools samples
- family control subject: family control unaffected subject
  Interventions: Genetic: genetic analysis; Biological: blood and stools samples

INTERVENTIONS:
Genetic: genetic analysis — genetic (Whole Exome Sequencing )
Biological: blood and stools samples — biological collection

SUMMARY:
This study highlight genetics mutations with major effect in Crohn's Disease (CD) by WES in individuals affected and healthy individuals from EPIMAD Inserm InVS registry families.

DETAILED DESCRIPTION:
The EPIMAD Registry covers a large area of Northern France (9 millions inhabitants) and collects all incident CD cases and data from CD multiplex families (families with 3 or more CD affected patients) in the Nord the Pas de Calais the Somme and the Seine Maritime. If the investigators could demonstrate that most CD cases from multiplex families were related to high frequency of NOD2 gene mutations, the investigators found some CD multiplex families without any NOD2 gene involvement. Thus in these families high prevalence of CD cases may rely on other major genetic susceptibility variant(s) that remain to be determined.

this clinical research Whole Exome Sequencing protocol, aiming to highlight genetics mutations with major effect in CD has been initiated.

This study is a familial genetic study with intra-familial controls. The genetics analyses are:

* Ascertain of no significant NOD2 mutation in the family members by Sanger DNA sequencing
* WES (CD patients and family controls unaffected subjects)
* Genotyping of all mutations found, case control and segregation analyses to validate their implication in CD.

ELIGIBILITY:
Inclusion Criteria:

* Crohn disease subject
* EPIMAD family with, at least, 3 Crohn disease subjects

Exclusion Criteria:

* Pregnant or lactating women

Ages: 5 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Crohn disease subject
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
NOD2 gene status | 8 months after recruiting
  One of the main inclusion criteria is the absence in the family (and thus in the proband) of any NOD2 mutation that could be related with the high occurrence of Crohn's Disease in the family. So verification of the lack of CD related NOD2 gene mutation is a prerequisite to the inclusion of the family in the protocol. This is achieved by Sanger sequencing of all exons, exon-intron junctions and search for already described intronic mutations in the family proband.

SECONDARY OUTCOMES:
Whole Exome Sequencing | 10 months after recruiting
  Whole Exome Sequencing will be performed in every subject from all families. All genetic variants will be filtered with bioinformatic tools. Genetic variants with putative biological effect, presents in affected CD patients and absents in their unaffected relatives will be further investigated (i.e. cosegregation with the disease, involvement in a given pathway....). This study remains a "pilot study" to identify genetic variants that may be involved in Crohn's Disease.

CONTACTS AND LOCATIONS:
Overall Officials: Corinne Gower, MD, PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- CHRU, Hôpital Claude Huriez, Lille, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Frade-Proud'Hon-Clerc S, Smol T, Frenois F, Sand O, Vaillant E, Dhennin V, Bonnefond A, Froguel P, Fumery M, Guillon-Dellac N, Gower-Rousseau C, Vasseur F. A Novel Rare Missense Variation of the NOD2 Gene: Evidencesof Implication in Crohn's Disease. Int J Mol Sci. 2019 Feb 15;20(4):835. doi: 10.3390/ijms20040835. PMID 30769939